CLINICAL TRIAL: NCT00086203
Title: Study of Talabostat and Rituximab in Advanced Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Point Therapeutics (Industry)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTH-203; FD-R-003021-01
Record Dates: First submitted 2004-06-28; First posted 2004-06-29 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2006-08

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — PT-100 dipeptide; talabostat; Tablets; Rituximab

INTERVENTIONS:
Drug: Talabostat mesylate (PT-100) tablets
Drug: Rituximab

SUMMARY:
The objective of this study is to assess the efficacy and safety of talabostat and rituximab in patients with advanced CLL who failed to respond, or have progressed following a prior response, to a fludarabine regimen.

DETAILED DESCRIPTION:
Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
INCLUSION CRITERIA:

* Men or women ≥18 years of age
* Histopathologically confirmed diagnosis of B-CLL expressing surface CD20 of any detectable intensity
* Rai Stage III or IV. Rai Stages I and II with massive or progressive lymphadenopathy or hepatosplenomegaly.
* Primary resistance to a fludarabine regimen (no PR or CR) or progressive disease within 1 year of a prior response
* ECOG performance status 0, 1, or 2
* Written informed consent

EXCLUSION CRITERIA:

* Therapy for CLL within 4 weeks of Study Day 1 (including chemotherapy, radiation, immunotherapy, cytokine or biologic [with the exception of hematopoietic growth factors]). Patients must have recovered from the adverse effects of prior therapy.
* Known primary or secondary malignancy of the central nervous system
* Any malignancy within the 5 years immediately prior to the first dose of study medication with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix
* Serum creatinine >2.0mg/dL (>176 micromol/L)
* AST or ALT ≥3 x the upper limit of normal (ULN)
* Total bilirubin ≥1.5 x ULN (unless secondary to Gilbert's)
* Positive serology for hepatitis B (HBsAg) or hepatitis C (anti-HCV antibody)
* Known positivity for HIV
* Prior organ allograft
* Concurrent comorbid medical conditions that, in the opinion of the investigator, preclude the safe delivery of the experimental treatment
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2007-09

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Ocala Oncology Center, Ocala, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Indiana Oncology/Hematology Consultants, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hematology/Oncology Centers of the Northern Rockies, Billings, Montana
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Queens Medical Associates, PC, Fresh Meadows, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU Medical Center, New York, New York
  - James P. Wilmot Cancer Center/University of Rochester, Rochester, New York
  - Raleigh Hematology/Oncology Clinic, Cary, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cancer Care Associates/Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Care Associates--Tulsa, Tulsa, Oklahoma
  - Cancer Centers of the Carolinas, Seneca, South Carolina
  - Texas Cancer Center/Abilene, Abilene, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates-Lake Wright Cancer Center, Norfolk, Virginia